CLINICAL TRIAL: NCT05848310
Title: Preoperative Serum FGF19 in the Prognosis of Biliary Atresia
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: SFPBA
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Biliary Atresia; Prognosis
Keywords: Biliary Atresia; FGF19
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Preoperative serum of biliary atresia patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Good prognosis + Poor prognosis: Good prognosis: the serum total bilirubin level was less than 20 umol/l three months after surgery, and no liver transplantation or death occurred within a year after surgery.
  Poor prognosis: the serum total bilirubin level was higher than 20 umol/l three months after surgery, and no liver transplantation or death occurred within a year after surgery.

SUMMARY:
To investigate the role of preoperative serum FGF19 level in the prognosis of biliary atresia.

DETAILED DESCRIPTION:
Kasai portoenterostomy is currently one of the main treatment methods for biliary atresia, but about 30% of children still require liver transplantation even after receiving the surgery. Accurate prognosis will help select the most suitable treatment method for children, but there is currently a lack of effective preoperative predictive indicators. Serum FGF19 has recently been considered a possible preoperative predictive indicator for biliary atresia, but its predictive value has not been confirmed in a large sample and in Asian population, thus the investigators try to further explore the prognostic value of serum FGF19 in children with biliary atresia based on a large sample.

ELIGIBILITY:
Inclusion Criteria:

* Samples diagnosed as biliary atresia in Children's Hospital of Fudan University
* Samples with one-year follow-up records after surgery
* Samples with a record of serum total bilirubin levels three months after surgery
* Samples with preoperative serum left（volume > 500ul)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study enrolled patients meeting following conditions.
  * Patients diagnosed as biliary atresia in Children's Hospital of Fudan University
  * Patients with at least one-year follow-up records after surgery
  * Patients with a record of serum total bilirubin levels three months after surgery
  * Patients with preoperative serum left（volume > 500ul)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Serum total bilirubin level (umol/l) | Three months after surgery
  The difference of serum total bilirubin level will be measured with ELISA( Enzyme Linked ImmunoSorbent Assay) three months after surgery
Native liver survival (%) | One year after surgery
  The difference of native liver survival will be measured according to the follow-up statue one year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No